CLINICAL TRIAL: NCT05394337
Title: Neoadjuvant PD-1 Plus TIGIT Blockade in Patients With Cisplatin-Ineligible Operable High-Risk Urothelial Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0928; NCI-2022-04565 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Malignancy
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atezolizumab (Experimental): Atezolizumab will be administered at a fixed dose of 1200 mg Q3W (1200 mg on Day 1 of each 21 day cycle),
  Interventions: Drug: Atezolizumab
- Tiragolumab (Experimental): Tiragolumab will be administered at a fixed dose of 600 mg intravenously Q3W on Day 1 of each 21-day cycle.
  Interventions: Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Given by vein (IV)
  Other Names: MPDL3280A; TECENTRIQ
  Arms: Atezolizumab
Drug: Tiragolumab — Given by vein (IV)
  Arms: Tiragolumab

SUMMARY:
To learn if the combination of atezolizumab and tiragolumab can help to control bladder cancer when it is given before surgery to remove the bladder and tumor.

DETAILED DESCRIPTION:
Primary Safety Objective:

•To evaluate the safety and tolerability oftiragolumab and atezolizumab in patients with muscle-invasive, high-risk UC who are ineligible for neoadjuvant cisplatin-containing chemotherapies.

Secondary Efficacy Objectives:

* To evaluate pathologic T0 rate after neoadjuvant treatment with tiragolumab and atezolizumab in patients with muscle-invasive, high-risk UC comparing to historical data (about 10% in patients with high-risk disease).
* To evaluate relapse-free survival (RFS) and overall survival (OS).

Exploratory Biomarker Objective :

• To assess immunologic/molecular responses to tiragolumab and atezolizumab in patients with muscleinvasive, high-risk UC who are ineligible for neoadjuvant cisplatin-containing chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age >18 years at time of signing Informed Consent Form
3. Ability to comply with the study protocol
4. Histologically or cytologically confirmed proof of muscle invasive urothelial cancer. This may include any patient requiring cystectomy (or nephroureterectomy to resect tumors), including muscle invasive disease (cT2-4aN0M0). Patients with the following high-risk features who are not candidates for traditional neoadjuvant chemotherapy will be included for this trial: micropapillary, sarcomatoid and plasmacytoid features; 3-D mass on exam under anesthesia (EUA); lymphovascular invasion; hydronephrosis (unless in the opinion of the treating physician, this is not due to tumor); high grade (grade 3) tumors of the ureter, renal pelvis, or tumors in these areas with radiographic abnormality large enough to recognize as an abnormal mass by CT or MRI imaging5; direct invasion of the prostatic stroma or the vaginal wall (i.e. cT4a disease). For patients in whom eligibility is unclear, final arbitration will be determined by the Principal Investigator.
5. Subjects must be considered cisplatin ineligible as per treating physician (Eastern Cooperative Oncology Group performance status (ECOG-PS) 2, creatinine clearance (CrCl) <60 mL/min, grade > 2 hearing loss, grade > 2 neuropathy, or New York Heart Association (NYHA) class III heart failure. See FDA draft guidance n adjuvant therapy in bladder cancer https://www.fda.gov/media/142544/download) or have refused cisplatinbased chemotherapy as a neoadjuvant therapy.
6. Tissue resected by transurethral resection of bladder tissue (TURBT) at the MD Anderson Cancer Center; if completed TURBT at the outside facility, it must be within three months and must transfer outside TURBT tumor tissues to MD Anderson for correlative research on this trial.
7. Eligible for R0 resection with curative intent at the time of screening, as confirmed by the operating attending surgeon and involved medical oncologist prior to study enrollment
8. Adequate pulmonary function to be eligible for surgical resection with curative intent, as assessed by PFTs performed within 6 months of planned resection and repeated at screening, if clinically indicated, including lung volumes, spirometry, and a diffusion capacity; and meeting at least one of the following criteria:

   1. Predicted postoperative (ppo) forced expiratory volume in 1 second (FEV1) and ppo diffusion capacity of the lung for carbon monoxide (DLCO) >40%
   2. Maximal oxygen consumption (VO2max) >15 mL/kg/min
9. If either ppoFEV1 or ppoDLCO is <40% or a pneumonectomy is planned, cardiopulmonary exercise testing must be performed and VO2max >15 mL/kg/min.
10. If PFTs were performed before 6 months of planned resection or have not been previously performed, they must be performed during the screening period.
11. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
12. Normal life expectancy, excluding lung cancer mortality risk
13. Adequate hematologic and -end organ and marrow function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

    1. ANC > 1.5 x 109

       /L (1500/µL) without granulocyte colony-stimulating factor support
    2. Lymphocyte count >0.5 x 109

       /L (500/µL)
    3. Platelet count >100 x109

       /L (100,000/µL) without transfusion
    4. Hemoglobin >90 g/L (9 g/dL)

1. Patients may be transfused to meet this criterion. e. AST, ALT, and ALP <2.5 x upper limit of normal (ULN) f. Total bilirubin <1.5 xULN with the following exception: Patients with known Gilbert disease (>3 xULN): who must have a baseline total bilirubin <3.0 mg/dL g. Creatinine clearance >45 mL/min (calculated using the Cockcroft-Gault formula) h. Serum albumin >25 g/L (2.5 g/dL)

14. For patients not receiving therapeutic anticoagulation: INR and aPTT <1.5 xULN

15. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen

16. Negative HIV test at screening

17. Negative hepatitis B surface antigen (HBsAg) test at screening

18. Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

a. Negative total hepatitis B core antibody (HBcAb) b. Positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA< 500 IU/mL. The HBV DNA test will be performed only for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test. c. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.

19. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs, as defined below:

a. Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for up to 23 weeks after the last dose of study drugs dose. Women must refrain from donating eggs during this same period. b. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (>12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations. c. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

d. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form. e. Women who would like to become pregnant after study treatment discontinuation should seek advice on oocyte cryopreservation prior to initiation of study treatment.

20. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

1. With a female partner of childbearing potential, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period, for up to 90 days after the final dose of the study drugs. Men must refrain from donating sperm during this same period.
2. With a pregnant female partner, men must remain abstinent or use a condom during the treatment period for 90 days after the final dose of the study drugs to avoid exposing the embryo.
3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
4. Men who would like to father a child after study treatment initiation should be advised regarding the conservation of sperm prior to treatment because of the possibility of irreversible infertility resulting from drugs used in this study.

Exclusion Criteria:

1. Illness or condition that may interfere with a patient's capacity to understand, follow, and/or comply with study procedures
2. Any prior therapy for urothelial cancer, including immunotherapy, chemotherapy, or radiotherapy
3. History of leptomeningeal disease
4. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 4 for a more comprehensive list of autoimmune diseases and immune deficiencies), with the exceptions listed below.

   1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

   i. Rash must cover <10% of body surface area ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
5. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
6. Active tuberculosis
7. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
8. Major surgical procedure, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
9. History of malignancy other than urothelial cancer within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
10. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion of the investigator, could impact patient safety
11. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment

    a. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
12. Prior allogeneic stem cell or solid organ transplantation
13. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
14. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment, within 90 days after the final dose of tiragolumab, or within 5 months after the final dose of atezolizumab
15. Current treatment with anti-viral therapy for HBV
16. Positive Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test at screening

    a. An EBV PCR test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.
17. Treatment with investigational therapy within 42 days prior to initiation of study treatment
18. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, anti-TIGIT, and anti-PD-L1 therapeutic antibodies.
19. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
20. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor- [TNF-] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    1. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after IND Medical Monitor confirmation has been obtained
    2. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose (< 10mg prednisone equivalent per day) corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
21. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
22. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation.
23. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment, within 90 days after the final dose of tiragolumab, 5 months after the final dose of atezolizumab. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate relapse-free survival (RFS) | Through study completion, an average of 1 year
To evaluate overall survival (OS). | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Padmanee Sharma, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org